CLINICAL TRIAL: NCT00796783
Title: A Study to Confirm the Presence of Recurrent or Persistent Cushing's Syndrome in Patients With Clinical Signs or Symptoms of Hypercortisolemia Who Have Been Treated for Cushing's Disease
Brief Title: A Study to Confirm Recurrent or Persistent Cushing's Syndrome in Patients With Signs or Symptoms of Hypercortisolemia
Status: Terminated | Type: Observational
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: C-1073-410
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's Disease; Cushing's Syndrome; Cushings; Pituitary; ACTH; Adrenocorticotropic hormone; Ectopic; Adrenal adenoma; Adrenal carcinoma; Adrenal autonomy; Cortisol; Hypercortisolemia; Cushinoid; Moon facies; Dorsalcervical fat; Plethora; Hirsutism; Violaceous striae; Hormone; Contraceptive; Endocrine; Cushing Syndrome; Ectopic ACTH Secretion
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; Pituitary Diseases; Choristoma; ACTH Syndrome, Ectopic; Adrenal Cortex Neoplasms; Hirsutism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with presumed Cushing's disease who have failed pituitary surgery and/or radiation and require medical treatment for recurrent or persistent Cushing's syndrome.
  Interventions: Drug: Cushing's syndrome confirmation

INTERVENTIONS:
Drug: Cushing's syndrome confirmation
  Other Names: Provide access to standard test procedures.

SUMMARY:
This is an observational study to confirm the presence of recurrent or persistent endogenous Cushing's syndrome in patients who have had primary surgical and/or radiation therapy for Cushing's disease and continue to manifest symptoms and signs of hypercortisolemia.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years of age.
* Have a presumptive diagnosis of Cushing's disease (Cushing's syndrome due to an ACTH secreting pituitary tumor).
* Have previously had pituitary surgery and/or pituitary radiation with the intent of curing or treating Cushing's disease.
* Have clinical symptoms and signs of hypercortisolism.
* Are able to provide written informed consent.
* Are expected to complete the study.

Exclusion Criteria:

* Are surgical candidates for pituitary surgery or have had pituitary surgery within 8 weeks before screening.
* Have taken any medication that may interfere with protocol testing procedures within 30 days of initial screening (phenobarbital, phenytoin, carbamazepine, oxcarabazepine, primidone, rifampin, rifapentine, rifabutin, ethosuximide, pioglitazone, efavirenz, neviparine, modafinil, St. Johns wort, glucorticoids, estrogen containing oral contraceptives).
* Have received investigational treatment (drug, biologic agent or device) within 30 days of screening.
* Have a non-endogenous source of hypercortisolemia such as factitious hypercortisolemia (exogenous source of glucocorticoid, iatrogenic Cushing's syndrome), factitious or therapeutic use of ACTH.
* Have Pseudo-Cushing's syndrome. Subjects with suspected Pseudo-Cushing's syndrome such as those with severe obesity, major depression or a history of alcoholism.
* Uncontrolled, clinically significant hypothyroidism or hyperthyroidism.
* Have renal failure as defined by a serum creatinine of 202 mg/dL.
* Elevated total bilirubin (>1.5x ULN), elevated ALT(>3x ULN) or AST (>3x ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presumed Cushing's disease who have failed pituitary surgery and/or radiation and require adjuvant medical treatment for recurrent or persistent Cushing's syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To confirm the presence of recurrent or persistent endogenous Cushing's syndrome in patients who have had primary surgical and/or radiation therapy for Cushing's disease and continue to manifest symptoms and signs of hypercortisolemia. | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Coleman Gross, MD, Study Director — Corcept Therapeutics
Locations (3):
- United States (3):
  - AMCR Institute Inc., Escondido, California
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Diabetes and Glandular Disease Research, San Antonio, Texas